CLINICAL TRIAL: NCT01927146
Title: Retrospective Study of Lauren Classifications and HER2 Status in Chinese Patients With Resectable Gastric Adenocarcinoma
Brief Title: Lauren Classifications and HER2 Status in Gastric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Vice president, Sun Yat-sen University
Other Study IDs: HER2 and Lauren
Record Dates: First submitted 2013-08-19; First posted 2013-08-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Gastric Cancer
Keywords: Lauren classification; HER2 status; Resectable gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Resectable gastric cancer: No intervention

SUMMARY:
By literature review, there is a clear trend towards a potential role for human epidermal growth factor receptor 2 (HER2) as a negative prognostic factor in gastric cancer was shown, but only in half of the analyses used multivariate statistics. Besides, For the studies in the current review that have looked at the Lauren classification in relation to HER2, a higher level of overexpression or amplification was found in the intestinal phenotype compared to the diffuse or mixed types. As lauren classification was reported as an independent prognostic factor result in favored outcomes in gastric cancer (GC), there may probably be histologic bias exists when compare overall survival (OS) between HER2 statuses without controlling this confounding. Similarly, patients with different disease settings (early stage and advanced stage; resectable and metastatic) affect outcomes either.

In this study, the investigators will retrospectively analyze HER2 status and lauren classification in 800 gastric patients who received gastrectomy in the Cancer Center of Sun Yat-Sen University between January 1996 and December 2006 with formalin-fixed and paraffin- embedded tumor tissue samples. To avoid potential influence by histologic classifications and disease settings, the investigators assess difference in OS between HER2 positive and HER2 negative groups in resectable Lauren classification of GCs, and further evaluate the prognostic value of HER2 status according to tumor-node-metastasis (TNM) stages.

DETAILED DESCRIPTION:
It's a single site, retrospective study by review of medical records and tissue testing.

Eight hundred gastric adenocarcinoma patients with integrity medical record and regular survival follow up who received gastrectomy in the Cancer Center of Sun Yat-Sen University between January 1996 to December 2006 were retrospectively studied.

Formalin-fixed and paraffin-embedded tumor tissue samples were retrospectively tested by human epidermal growth factor receptor 2 (HER2) and Lauren classification status. Her2 positive was defined as: immunohistochemistry (IHC) 2+ and fluorescence in situ hybridization (FISH) +; or IHC 3+.

1. After HER2 status and lauren classification identifying, population used in overall survival (OS) comparison between Cohort 1(HER2 positive) and Cohort 2 (negative group) were carried out. According to Tumor-node-metastasis (TNM) classification, OS were to be compared between cohorts by different stages.
2. Correlate histopathological characteristics with HER2 status and lauren classification were performed in the total 800 patients. Meanwhile, independent prognostic factors identification was to be confirmed in clinicopathological features, including gender (male or female), age at diagnosis, tumor size (≤5cm or >5cm), location of primary tumor (proximal or distal), histology subtypes (well + moderate differentiated adenocarcinoma or poorly + signet ring cell differentiated adenocarcinoma), lauren classifications (diffuse type or intestinal type or mixed type), anemia (yes or no), angiolymphatic invasion (yes or no), the TNM staging system (American Joint Committee on Cancer (AJCC) 7th edition), and HER2 status (negative and positive).

ELIGIBILITY:
Inclusion Criteria:

1. Patients' admission date: 1996-2006.
2. Histologically confirmed gastric adenocarcinoma patients and underwent gastrectomy.
3. Adequate paraffin- embedded tumor tissue sample for pathologic and human epidermal growth factor receptor 2 (HER2) status analysis.
4. Integrity medical records with regular survival follow up, the overall survival (OS) could be sourced.

Exclusion Criteria:

1. Age<18 years old.
2. Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is single site, retrospective study by review of medical records and tissue testing.
  800 gastric adenocarcinoma patients with integrity medical record and regular survival follow up who received gastrectomy in the Cancer Center of Sun Yat-Sen University between January 1996 to December 2006 were retrospectively studied.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At least 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Qiu M, Zhou Y, Zhang X, Wang Z, Wang F, Shao J, Lu J, Jin Y, Wei X, Zhang D, Wang F, Li Y, Yang D, Xu R. Lauren classification combined with HER2 status is a better prognostic factor in Chinese gastric cancer patients. BMC Cancer. 2014 Nov 7;14:823. doi: 10.1186/1471-2407-14-823. PMID 25380654